CLINICAL TRIAL: NCT01590056
Title: Mapping and Manipulating the Motor, Emotional and Cognitive Territories of the Subthalamic Area in Deep Brain Stimulation Treated Parkinson Patients
Brief Title: Emotional and Cognitive Subthalamic Nucleus in Deep Brain Stimulation Treated Parkinson Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Renana Eitan, Head, Neuropsychiatry Clinic, Hadassah Medical Organization
Other Study IDs: STN_Cog_HMO-CTIL; 0064-12-HMO (Other: HMO)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Parkinson's Disease
Keywords: Mapping limbic areas of the STN; neuronal responses to stimuli during surgery
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PD patients: PD patients that are treated or are candidates for treatment with STN DBS
  Interventions: Other: Electrophysiological recording

INTERVENTIONS:
Other: Electrophysiological recording — During the surgery for bilateral DBS electrode implantation, electrophysiological recording from the STN will be made while patients are:
  1. listening to nonverbal affect bursts corresponding to emotions
  2. applying a simple go-no-go auditory test

SUMMARY:
About 300 patients with Parkinson's disease (PD) have been successfully treated by deep brain stimulation (DBS) during the last 10 years in Hadassah. In most of the patients the site of stimulation is the subthalamic nucleus (STN). Recent studies by our group and others have demonstrated that the STN is divided into motor and non-motor areas. The investigators have recently shown that electrophysiological mapping of the STN during the surgery can differentiate motor and non-motor areas of the STN. Existing methods of adjustment of DBS parameters aim at amelioration of the motor signs and therefore with inactivation of the STN motor territory only. Although the DBS parameter setting is believed to influence the mental and cognitive states, there is no data that correlates stimulation parameters with mental and cognitive state. In addition, DBS parameter setting is also believed to influence important verbal functions which are partially related to motor, mental and cognitive states, but no data correlates the verbal function with the DBS stimulation parameters.

The investigators hypothesize that the cognitive areas of the STN have distinct electrophysiological properties similar to our findings with the limbic / mental areas of the STN. The investigators further hypothesize that specific stimulation of these cognitive areas can influence the cognitive state and thus treatment with cognitive-adjusted DBS can improve the cognitive symptoms of PD.

In this project, the investigators intend to map the motor, emotional and cognitive areas of the STN using neuronal (single units) responses to emotional voices and cognitive tasks and to identify the emotional and cognitive spectral signature of the STN single unit activity using spectral analysis and neuronal responses to emotional voices and cognitive tasks. In addition the investigators intend to find the neuronal signature of speech and to find the correlation between motor, mental and limbic electrophysiology to speech. The investigators also intend to investigate the motor, emotional and cognitive processing of PD patients by manipulating the stimulation of the STN. The proposed study will combine neural recording, stimulation and psychological and cognitive tests to shed new light on processing in the basal ganglia, as well as to provide better treatment for PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically definite PD treated / candidates for treatment with DBS (patients with advanced idiopathic PD who are deemed appropriate for DBS surgery).
* Patients will be included in the study irrespective of whether a diagnosis of major depression (mild to moderate but not severe MDD) is fulfilled at baseline. Patients without depression will be monitored in the study for evidence of treatment emergent depression. Patients with depression will be monitored for antidepressant effects of stimulation change.
* Age 40-75 years
* Male or female.
* Competent and willing to give written informed consent.

Exclusion Criteria:

* Significant suicidal risk [Hamilton Depression scale item 3 (suicide) >2].
* Comorbidity with any Psychotic Disorder, Bipolar Disorder, Post Traumatic Stress Disorder (PTSD), Eating Disorder.
* Lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months
* Significant cognitive decline, as measured by Addenbrooke's Cognitive Examination (ACE) and the Frontal Assessment Battery (FAB).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients that are treated or are candidates for treatment with STN DBS will be followed for 12 months (n=20). These patients will represent a consecutive sample of community based PD patients who will be enrolled in a prospective, open label, clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Mapping the motor, emotional and cognitive areas of the STN using neuronal (single units) responses to motor stimuli, emotional voices and cognitive tests during surgery. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renana Eitan, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel